CLINICAL TRIAL: NCT05085405
Title: Anticoagulation With Enhanced Gastrointestinal Safety (AEGIS): A Pilot Trial to Evaluate Clinician- and Patient-facing Strategies to Reduce Upper Gastrointestinal Bleeding Risk in Patients on Combination Antithrombotic Therapy
Brief Title: Anticoagulation With Enhanced Gastrointestinal Safety (AEGIS) Trial
Acronym: AEGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jacob E Kurlander, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00201535; K23DK118179 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: combination antithrombotic therapy; proton pump inhibitor; peptic ulcer disease; gastroprotection; warfarin; anticoagulation; patient safety
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Peptic Ulcer

STUDY DESIGN:
Intervention Model Description: Assignment to one of two clinician-level implementation strategies will be done at the cluster level according to the identity of the clinician to be contacted. Clinicians will be randomized 1:1 to receive either clinician notification (CN) or clinician notification + nurse facilitation (CN+NF). Patients within each clinician cluster will also be individually randomized to receive a patient activation guide or to a usual care arm.
  There are 2 arms for each group (patients and clinicians).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinician Notification only (Experimental)
  Interventions: Behavioral: Clinician notification
- Clinician Notification with Nurse Facilitation only (Experimental)
  Interventions: Behavioral: Clinician Notification with Nurse Facilitation
- Clinician Notification / Patient Activation (Experimental)
  Interventions: Behavioral: Clinician Notification / Patient Activation
- Clinician Notification with Nurse Facilitation / Patient Activation (Experimental)
  Interventions: Behavioral: Clinician Notification with Nurse Facilitation / Patient Activation

INTERVENTIONS:
Behavioral: Clinician notification — An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
  In this arm, patients receive no additional interventions beyond that provided during treatment as usual.
  Arms: Clinician Notification only
Behavioral: Clinician Notification with Nurse Facilitation — An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
  In this arm, patients receive no additional interventions beyond that provided during treatment as usual.
  Arms: Clinician Notification with Nurse Facilitation only
Behavioral: Clinician Notification / Patient Activation — An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
  Patient Activation:
  An anticoagulation clinic nurse sends the patient an 8-page written guide, either through the patient portal or by mail. The guide provides education on upper GI bleeding risk and encourages patients to talk with their clinician about medication changes to reduce their bleeding risk.
  Arms: Clinician Notification / Patient Activation
Behavioral: Clinician Notification with Nurse Facilitation / Patient Activation — An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
  Patient Activation:
  An anticoagulation clinic nurse sends the patient an 8-page written guide, either through the patient portal or by mail. The guide provides education on upper GI bleeding risk and encourages patients to talk with their clinician about medication changes to reduce their bleeding risk.
  Arms: Clinician Notification with Nurse Facilitation / Patient Activation

SUMMARY:
This is a pragmatic, single center, feasibility pilot cluster randomized trial with embedded individual randomization to evaluate implementation strategies to increase the use of evidence-based practices to reduce upper gastrointestinal bleeding risk in patients using combination antithrombotic therapy (including warfarin) and that are managed by the Michigan Medicine anticoagulation monitoring service.

DETAILED DESCRIPTION:
In February 2022, the IRB approved adding a small additional substudy for the collection of exploratory qualitative outcomes only, involving up to 8 primary care physicians. As no data for the primary and secondary outcome measures was collected for this substudy, and all data collection for this group was related to exploratory outcome measures and collected through qualitative interviews with clinicians, no inclusion exclusion criteria specific to the participants in this substudy are listed, nor does the data collection from them show in the study completion date or results data. However, these physicians (n=8) and their patients (n=9) are counted in the actual enrollment total since they were randomized to intervention arms and received study interventions.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Enrollment with the Michigan Medicine anticoagulation monitoring service
* Currently prescribed warfarin with anticipated use for greater or equal to 90 days on day 1 of trial enrollment, according to electronic medical record documentation
* Currently prescribed an antiplatelet drug (aspirin, clopidogrel, ticagrelor, or prasugrel) according to the electronic medical record medication list

Exclusion Criteria for Patients:

* Prescribed a Proton Pump Inhibitor (PPI)
* Documented intolerance or allergy to PPI use
* Left ventricular assist device
* Heart transplant

Inclusion Criteria for Clinicians:

* Practicing cardiologists at Michigan Medicine who in the prior year had a face-to-face or virtual visit with a patient who meets eligibility criteria for this study
* Practicing clinicians in any specialty who are designated as the clinician of record with the anticoagulation clinic for a patient who meets eligibility criteria

Exclusion Criteria for Clinicians:

- Cardiologists specializing in electrophysiology unless they are the clinician of record for a patient followed by the anticoagulation service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kurlander, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurlander JE, Helminski D, Lanham M, Henstock JL, Kidwell KM, Krein SL, Saini SD, Richardson CR, De Vries R, Resnicow K, Ruff AL, Wallace DM, Jones EK, Perry LK, Parsons J, Ha N, Alexandris-Souphis T, Dedrick D, Aldridge E, Barnes GD. Development of a multicomponent implementation strategy to reduce upper gastrointestinal bleeding risk in patients using warfarin and antiplatelet therapy, and protocol for a pragmatic multilevel randomized factorial pilot implementation trial. Implement Sci Commun. 2022 Jan 28;3(1):8. doi: 10.1186/s43058-022-00256-8. PMID 35090577

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Clinicians (n=8) and patients (n=9) in the PCP substudy did not undergo data collection for the primary or secondary outcome measures. Clinician participants were invited by email to participate in semi-structured qualitative interviews for exploratory outcome measures. Review of patient charts occurred at week 5 solely to ascertain whether the clinician responded to the clinician-facing intervention to inform clinician interviews, but no additional chart review or patient assessments were done.
Groups:
- Patient Arm - Clinician Notification Only: Clinician notification: An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
  In this arm, patients receive no additional interventions beyond that provided during treatment as usual.
- Patient Arm - Clinician Notification With Nurse Facilitation Only: Clinician Notification with Nurse Facilitation: An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
  In this arm, patients receive no additional interventions beyond that provided during treatment as usual.
- Patient Arm - Clinician Notification / Patient Activation: Clinician Notification / Patient Activation: An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
  Patient Activation:
  An anticoagulation clinic nurse sends the patient an 8-page written guide, either through the patient portal or by mail. The guide provides education on upper GI bleeding risk and encourages patients to talk with their clinician about medication changes to reduce their bleeding risk.
- Patient Arm - Clinician Notification With Nurse Facilitation / Patient Activation: Clinician Notification with Nurse Facilitation / Patient Activation: An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
  Patient Activation:
  An anticoagulation clinic nurse sends the patient an 8-page written guide, either through the patient portal or by mail. The guide provides education on upper GI bleeding risk and encourages patients to talk with their clinician about medication changes to reduce their bleeding risk.
- Clinician Arm - Notification Only: Clinician notification: An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
- Clinician Arm - Notification With Nurse Facilitation: Clinician Notification with Nurse Facilitation: An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
Period: Overall Study
Arm/Group | Patient Arm - Clinician Notification Only | Patient Arm - Clinician Notification With Nurse Facilitation Only | Patient Arm - Clinician Notification / Patient Activation | Patient Arm - Clinician Notification With Nurse Facilitation / Patient Activation | Clinician Arm - Notification Only | Clinician Arm - Notification With Nurse Facilitation
Started | 13 | 13 | 12 | 13 | 6 | 6
Completed (Patients were considered to have completed the overall study if they continued to meet all eligibility criteria at the time of study entry (e.g., not screen failures), and if they were still enrolled in the Anticoagulation Monitoring Service 5 weeks after study entry and eligible for the week 5 patient phone assessment per study protocol. Clinicians were considered to have completed the overall study if they received the clinician-level intervention for any of their eligible patients.) | 13 | 13 | 11 | 10 | 6 | 6
Not Completed | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Patient closed to the anticoagulation clinic monitoring service | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Patient started PPI prior to intervention delivery. | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per study protocol, patient participants who were randomized but no longer met eligibility criteria at the time of study entry (e.g., screen failures), and those who received the study interventions but discontinued warfarin therapy or unenrolled from the Anticoagulation Monitoring Service during the first 5 weeks of study participation were not included in the study analyses.
Groups:
- Clinician Arm - Clinician Notification: Clinician notification: An anticoagulation clinic nurse sends a templated letter to the patient's clinician and identifies the patient as high risk for upper GI bleeding, summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), provides a link to guidance on evidence-based use of antiplatelet therapy, and asks that the clinician manage any medication changes.
- Clinician Arm - Clinician Notification With Nurse Facilitation: Clinician Notification with Nurse Facilitation: An anticoagulation clinic nurse sends an individualized letter to the patient's clinician which identifies the patient as high risk for upper GI bleeding and summarizes options for medication optimization (e.g., discontinuation of antiplatelet therapy or initiation of a proton pump inhibitor for gastroprotection), but in addition includes a summary of the patient's history of atherosclerotic cardiovascular disease and a concise guidance summary on appropriate use of antiplatelet therapy for relevant indications. The anticoagulation nurse will assist with order entry for any new medications and also provide education on medication changes to the patient upon request by the clinician.
- Total: Total of all reporting groups
Arm/Group | Patient Arm - Clinician Notification Only | Patient Arm - Clinician Notification With Nurse Facilitation Only | Patient Arm - Clinician Notification / Patient Activation | Patient Arm - Clinician Notification With Nurse Facilitation / Patient Activation | Clinician Arm - Clinician Notification | Clinician Arm - Clinician Notification With Nurse Facilitation | Total
Number analyzed (Participants) | 13 | 13 | 11 | 10 | 6 | 6 | 59
Age, Customized [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    Age of Participants at Baseline: number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    Age of Participants at Baseline: Age 18-59 | 5 | 7 | 3 | 5 |  |  | 20
    Age of Participants at Baseline: Age 60-69 | 3 | 2 | 4 | 1 |  |  | 10
    Age of Participants at Baseline: Age 70-79 | 4 | 4 | 3 | 3 |  |  | 14
    Age of Participants at Baseline: Age 80+ | 1 | 0 | 1 | 1 |  |  | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 3 | 0 | 3 | 20
  Male | 6 | 10 | 7 | 7 | 6 | 3 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    Hispanic or Latino | 0 | 1 | 0 | 0 |  |  | 1
    Not Hispanic or Latino | 13 | 12 | 11 | 10 |  |  | 46
    Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    American Indian or Alaska Native | 0 | 0 | 0 | 0 |  |  | 0
    Asian | 0 | 1 | 0 | 1 |  |  | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  |  | 0
    Black or African American | 1 | 1 | 0 | 1 |  |  | 3
    White | 11 | 10 | 11 | 8 |  |  | 40
    More than one race | 0 | 0 | 0 | 0 |  |  | 0
    Unknown or Not Reported | 1 | 1 | 0 | 0 |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 11 | 10 | 6 | 6 | 47
Concomitant Medication - Oral Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    (all) | 1 | 0 | 0 | 0 |  |  | 1
Concomitant Medication - Selective Serotonin Reuptake Inhibitors (SSRIs) [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    (all) | 3 | 1 | 0 | 1 |  |  | 5
Concomitant Medication - Aldosterone Antagonists [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    (all) | 2 | 4 | 1 | 0 |  |  | 7
Concomitant Medication - Oral Glucocorticoids [Count of Participants; unit: Participants] — Population: This data was not collected for physician participants.
  Participants
    number analyzed (Participants) | 13 | 13 | 11 | 10 | 0 | 0 | 47
    (all) | 4 | 0 | 1 | 2 |  |  | 7
Clinician Specialty [Count of Participants; unit: Participants] — This measure applies only to Clinician participants. Population: This data was not collected for patient participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 12
    Cardiology |  |  |  |  | 3 | 3 | 6
    Surgery |  |  |  |  | 2 | 2 | 4
    Primary Care |  |  |  |  | 0 | 1 | 1
    Neurology |  |  |  |  | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Randomized Patients That Complete a Brief Medication Review Phone Call at Week 5
Description: The proportion of randomized patients that complete a brief medication review phone call at week 5 after up to 3 attempts.
Time Frame: Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Notification Only | Clinician Notification With Nurse Facilitation Only | Clinician Notification / Patient Activation | Clinician Notification With Nurse Facilitation / Patient Activation
Number analyzed (Participants) | 13 | 13 | 11 | 10
Participants | 7 | 12 | 8 | 8

2. Secondary Outcome: Feasibility of Delivering Intervention Components as Intended
Description: The proportion of patient participants that received all implementation components to which they were randomized in the appropriate time frame.
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Notification Only | Clinician Notification With Nurse Facilitation Only | Clinician Notification / Patient Activation | Clinician Notification With Nurse Facilitation / Patient Activation
Number analyzed (Participants) | 13 | 13 | 11 | 10
Participants | 13 | 13 | 11 | 10

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Description: Per protocol, this study did not proactively monitor for adverse events as the trial constituted a quality improvement effort intended to improve the use of evidence-based practices, and all decisions regarding changes in drug treatment were made by patients' own clinicians as part of usual care. However, if any adverse events were identified during data collection, the study team was instructed to document them in an adverse events database for regulatory review.
Arm/Group | Patient Arm - Clinician Notification Only | Patient Arm - Clinician Notification With Nurse Facilitation Only | Patient Arm - Clinician Notification / Patient Activation | Patient Arm - Clinician Notification With Nurse Facilitation / Patient Activation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT05085405/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT05085405/ICF_000.pdf